CLINICAL TRIAL: NCT03843437
Title: Lyocell as an Adjunct Treatment for Moderate to Severe Atopic Dermatitis in Children
Brief Title: Tencel vs. Standard Cotton Therapeutic Garments as an Adjunct Treatment for Moderate to Severe Atopic Dermatitis in Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study expired in IRB.
Sponsor: Johns Hopkins University (Other)
Collaborators: AD RescueWear (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00176371
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2021-09

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Tencel fabric; cotton fabric
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Fifty children age 6 months to 6 years with moderate to severe eczema will be recruited from the Johns Hopkins pediatric dermatology clinic and randomized (1:1) to be treated with Tencel vs. cotton therapeutic garments in addition to standard eczema care. Randomization will be computer-generated and parents will be blinded to whether the children receive Tencel vs. cotton garments.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Tencel Therapeutic Garments (Experimental): Children in this group will wear Tencel Therapeutic Garments
  Interventions: Device: Tencel Therapeutic Garments
- Cotton Therapeutic Garments (Placebo Comparator): Children in this group will wear Cotton Therapeutic Garments
  Interventions: Device: Cotton Therapeutic Garments

INTERVENTIONS:
Device: Tencel Therapeutic Garments — Children age 6 months to 3 years will wear a Tencel full body suit with feet and mittens, while children age 3-6 years will wear Tencel long-sleeve shirts and pants that do not cover the hands and feet. Children will wear the study garments at night but may also wear garments during the day if desired.
  Other Names: AD RescueWear "Rescue Suit"
  Arms: Tencel Therapeutic Garments
Device: Cotton Therapeutic Garments — Children age 6 months to 3 years will wear a cotton full body suit with feet and mittens, while children age 3-6 years will wear cotton long-sleeve shirts and pants that do not cover the hands and feet. Children will wear the study garments at night but may also wear garments during the day if desired.
  Arms: Cotton Therapeutic Garments

SUMMARY:
Approximately 15-20% of children in the United States suffer from the symptoms of atopic dermatitis (eczema), which include pruritus, pain, irritation, and difficulty sleeping. Tencel fabric has been marketed as a superior fabric for children with atopic dermatitis due to improved moisture absorption and decreased bacterial growth compared to cotton and synthetic fabrics. However, no dermatologic studies have been conducted on Tencel fabric. The investigators' objective is to perform a randomized double-blinded trial comparing Tencel garments to traditional cotton for children with moderate to severe atopic dermatitis. The investigators hypothesize that children in the Tencel group will demonstrate improvement in Eczema Area and Severity Index (EASI) scores, Investigator's Global Assessment, pruritus as measured by ItchyQoL: A Pruritus-Specific Quality of Life Instrument, and Children's Dermatology Life Quality Index (CDQLI) or Infant's Dermatitis Quality of Life Index (IDQoL).

An randomized double-blind trial of 12 weeks duration will be conducted. Fifty children age 6 months to 6 years with moderate to severe eczema will be recruited from the Johns Hopkins pediatric dermatology clinic and given 6 weeks of standard skin directed therapy followed by 6 weeks during which children will be randomized to treatment with Tencel vs. cotton therapeutic garments in addition to standard eczema care. The primary outcome will be eczema severity as assessed by EASI score by blinded and trained investigators. Secondary outcomes will include patient-reported eczema symptoms (assessed through quality of life and pruritus scales, CDQLI or IDQoL and ItchyQoL scores) and frequency of infection of eczema lesions. Adherence with wearing study garments and usage of standard eczema treatments (topical corticosteroids and calcineurin inhibitors, emollients, and wet/dry wraps) will also be assessed.

DETAILED DESCRIPTION:
Atopic dermatitis (eczema) is a chronically recurrent, pruritic disorder most common in infants and young children. It is one of the most common pediatric dermatologic disorders, affecting 15-20% of all children between 6 months and 10 years of age. The vast majority of affected children (up to 85%) have the first outbreak during infancy. The distribution of lesions is characteristically symmetric, involving the face and extensor surfaces during infancy and the flexural surfaces in later childhood. Afflicted children experience pruritic erythematous vesicles, papules, and plaques that weep and crust. Studies have found that up to 34% of children with atopic dermatitis report a "large or extremely large" effect on quality of life, and over 60% report experiencing sleeplessness due to itching and soreness. Other common frustrations include miserable mood changes, difficulties with dressing and bathing, and social isolation.

Traditionally, eczema guidelines have recommended loose cotton clothing and avoidance of rough fabrics such as wool which may cause irritation. Tencel is a botanic fiber derived from raw wood and has been marketed as a superior fabric for children with eczema. Industry studies of Tencel reported a 50% increase in moisture absorption compared to cotton and up to 2000 times less bacterial growth compared to polyamide (Tencel also had less bacterial growth than cotton or polyester). However, to date, no dermatologic studies have been conducted on the use of Tencel clothing to treat children with eczema. Because the investigators' department has observed several children achieve impressive reductions in eczema severity while using Tencel clothing, the investigators seek to conduct a formal study of this new textile.

A double blind randomized trial of 3 months duration will be conducted. Fifty children age 6 months to 6 years with moderate to severe eczema will be recruited from the Johns Hopkins pediatric dermatology clinic and randomized (1:1) to be treated with Tencel vs. cotton therapeutic garments in addition to standard eczema care. Randomization will be computer-generated and parents will be blinded to whether the children receive Tencel vs. cotton garments. Children will be stratified into age greater or less than 3 years. Children age 6 months to 3 years will wear either a Tencel or cotton full body suit with feet and mittens, while children age 3-6 years will wear Tencel or cotton long-sleeve shirts and pants that do not cover the hands and feet. Children will wear the study garments at night but may also wear garments during the day if desired (parent will estimate percentage of daytime hours that child wears garment). Parents will receive calendars and stickers to record nights that children wear the study garments, with a goal of wearing the study garments greater than 50% of the time. Blinded dermatology residents and fellows will assess EASI scores and Investigator's Global Assessment scores for each child at study initiation, 1 month, 2 months, and 3 months. CDQLI or IDQoL and ItchyQoL will also be assessed at each clinic visit. While some clinical photographs may be taken according to parental consent, no photographs will be taken of the genital area.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate or severe atopic dermatitis based on Eczema Area and Severity Index (EASI) score (moderate=6-22.9; severe=23-72)
* At least one active patch of atopic dermatitis at time of study
* Parent/guardian able to give informed consent

Exclusion Criteria:

* Systemic medication or oral steroids within past 3 months (includes light therapy),
* Started new atopic dermatitis treatment regimen within the past month,
* Using wet/dry wraps > once/week

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-04-28 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
Change in Atopic Dermatitis Severity score as assessed by Eczema Area and Severity Index (EASI) score | Baseline (At study initiation), 1 month, 2 months, and 3 months
  Assessment of erythema, excoriation, swelling, and lichenification on four body sites, scores range from 0-71. 0=clear, 0.1-5.9=mild, 6.0-22.9=moderate, 23.0-72=severe. A 3 point change in EASI score will be considered clinically significant for this study.
Change in Atopic Dermatitis Severity score as assessed by Investigator's Global Assessment for Atopic Dermatitis score | Baseline (At study initiation), 1 month, 2 months, and 3 months
  Physicians decide which of the following five categories best fits the patient:
  0 = clear: "No inflammatory signs of atopic dermatitis (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Post-inflammatory hyperpigmentation or hypopigmentation may be present."
  1. = almost clear: "Barely perceptible erythema, barely perceptible induration/papulation, and/or minimal lichenification. No oozing or crusting."
  2. = mild: "Slight but definite erythema (pink), slight but definite induration/papulation, and/or slight but definite lichenification. No oozing or crusting."
  3. = moderate: "Clearly perceptible erythema (dull red), clearly perceptible induration/papulation, and/or clearly perceptible lichenification. Oozing and crusting may be present."
  4. = severe: "Marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification. Disease is widespread in extent. Oozing or crusting may be present."

SECONDARY OUTCOMES:
Change in patient-reported pruritus as assessed by ItchyQoL | Baseline (At study initiation), 1 month, 2 months, and 3 months
  A Pruritus-Specific Quality of Life Instrument, assesses pruritus symptoms, resulting functional limitations, and patient emotions. Symptoms within the past 7 days are assessed, and scored 1 to 5 for both frequency (1=never, 5=all the time) and patient distress (1=not bothered, 5=severely bothered).
Change in patient-reported quality of life as assessed by Children's Dermatology Life Quality Index (CDQLI) | Baseline (At study initiation), 1 month, 2 months, and 3 months
  The most widely used instrument for measuring the impact of skin disease on quality of life (QOL) in children. Scores symptoms, embarrassment, friendships, clothes, playing, sports, school, bullying, sleep, and impact of treatment on 0 to 3. Scores of 0-1=no effect on QOL, 2-6=small effect, 7-12=moderate effect, 13-18=very large effect, and 19-30=extremely large effect. Validated for ages 4-16 years and available in text and cartoon versions.
Change in patient-reported quality of life as assessed by Infant's Dermatitis Quality of Life Index (IDQoL) | Baseline (At study initiation), 1 month, 2 months, and 3 months
  Designed for children age 0-3 years with atopic dermatitis. Parent/caregiver scores ten questions from 0-3 based on symptoms within the past week: itching and scratching, mood of the child, time to fall asleep, interference with playing/swimming/other activities, problems with mealtimes, problems during treatment, comfort with dressing, and problems with bathing. The maximum score is 30 and minimum is 0.
Incidence of superinfection of Atopic Dermatitis Lesions | 12 weeks
  The incidence of superinfection of atopic dermatitis lesions will be compared between the Tencel vs. cotton groups

CONTACTS AND LOCATIONS:
Overall Officials: Annie Grossberg, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Pediatric Dermatology Clinic, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No